CLINICAL TRIAL: NCT05747612
Title: Mental Coaching and Counseling for Bipolar Patients: Dealing With Moments of Crisis in
Brief Title: Mental Coaching and Counseling for Bipolar Patients: Dealing With Moments of Crisis in Times of COVID-19.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Principal Investigator, Mazza Marianna, Medical Doctor, Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 3275
Record Dates: First submitted 2023-02-26; First posted 2023-02-28 (Actual); Last update posted 2023-03-01 (Actual); Status verified 2023-02

CONDITIONS: To Determine the Incidence of Depression in Subjects Affected by Bipolar Disorder
MeSH Terms: interventions — Counseling

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with Bipolar Disorder (Other)
  Interventions: Other: Counseling and Coaching

INTERVENTIONS:
Other: Counseling and Coaching — Counseling is "the art of helping yourself", that is, a helping relationship based on a series of interventions and stimuli for creativity, aimed at pursuing and maintaining an ever better relational, social and existential quality of life. Coaching is a fundamentally action-oriented method, aimed at concrete changes, the improvement of performance and the achievement of objectives.

SUMMARY:
The goal of this interventional study is to evaluate some outcome parameters at the time of enrollment (T0), during the treatment (T1 and T2) and at the end (T3) of the subjects who will have carried out an individual counseling intervention or mental coaching. The aim is to determine the incidence of depression, trait anxiety, state anxiety, sleep disorders, resilience, defense mechanisms, distress caused by stressful events in a sample of subjects affected by Bipolar Disorder.

ELIGIBILITY:
Inclusion Criteria:

* Recruited subjects have a diagnosis of Bipolar Disorder and are 18 years of age or older.

Exclusion Criteria:

* Previous or current intellectual disability in accordance with the Diagnostic and Statistical Manual of Mental Disorders, DSM-5.
* Patients who are unable to express consent and who do not have a caregiver who can give it for them.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2022-01-25 (Actual); Study Completion 2023-02-01 (Actual)

PRIMARY OUTCOMES:
To determine the incidence of depression, trait anxiety, state anxiety, sleep disorders, resilience, defense mechanisms, distress caused by stressful events in a sample of subjects affected by Bipolar Disorder. | 12 months
  Administration of psychometric scales

SECONDARY OUTCOMES:
To ascertain the presence of evolutionary and maturational trends in the defensive structure especially in the face of a totally unpredictable and unexpected situation such as the COVID-19 pandemic. | 12 months
  Administration of psychometric scales

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione Policlinico Gemelli IRCCS, Rome, ROMA, Italy

IPD SHARING:
Plan to Share IPD: No